CLINICAL TRIAL: NCT07170150
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Study of Trontinemab in Participants With Early Symptomatic Alzheimer's Disease (MCI to Mild Dementia Due to AD)
Brief Title: A Clinical Trial of Trontinemab in Participants With Early Symptomatic Alzheimer's Disease
Acronym: TRONTIER 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN45447
Record Dates: First submitted 2025-09-10; First posted 2025-09-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Alzheimers Disease
Keywords: Early Alzheimers Disease; Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trontinemab (Experimental): Participants will receive intravenous (IV) trontinemab.
  Interventions: Drug: Trontinemab
- Placebo (Placebo Comparator): Participants will receive IV placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trontinemab — Participants will receive IV trontinemab
  Other Names: RO7126209
  Arms: Trontinemab
Other: Placebo — Participants will receive IV placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of trontinemab in participants with early symptomatic Alzheimer's disease (AD) (mild cognitive impairment [MCI] to mild dementia due to AD).

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to complete all aspects of the study (including MRI, clinical genotyping, and PET imaging or CSF as applicable) for the duration of the study. The participant should be capable of completing assessments either alone or with the help of the study partner
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eyewear and hearing aids are permitted)
* Evidence of AD pathological process, as confirmed on amyloid PET scan. A CSF tau181/Aβ42 ratio may be used as an alternative option if amyloid PET is not available
* Probable AD dementia or MCI due to AD, also known as an Alzheimer's clinical syndrome clinical Stage 3 or Stage 4
* Screening MMSE score ≥ 22 and CDR-GS of 0.5 or 1.0
* Participant- and/or Informant-reported history of cognitive decline with gradual onset and progression over the last 1 year before screening
* A Repeatable Battery for the Assessment of Neuropsychological Status Delayed Memory Index (RBANS DMI) score of 85 or order
* Availability of a "study partner" as defined by the protocol

Exclusion Criteria:

* Any evidence of a condition other than AD that may affect cognition
* History or presence of clinically significant cerebrovascular disease
* History of severe, clinically significant (persistent neurologic deficit or structural brain damage) central nervous system (CNS) trauma
* History or presence of clinically significant intracranial mass
* MRI evidence of significant cerebral abnormalities or inability to tolerate MRI procedures or contraindication to MRI
* Any other medical conditions (e.g., cardiovascular, hepatic, renal disease) which are not stable and adequately controlled or which in the opinion of the investigator could affect the participant's safety in the study or interfere with the study assessments
* History of malignancy with the following exceptions: if considered to be cured; malignancies with a negligible risk of metastasis or death

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-06-07 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 72 in Clinical Dementia Rating, Sum of Boxes (CDR-SB) | Baseline - Week 72

SECONDARY OUTCOMES:
Change from baseline through Week 72 in Alzheimer's Disease Assessment Scale-Cognition 13 (ADAS-Cog-13) | Baseline - Week 72
Change from baseline through Week 72 in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) total score and instrumental score | Baseline - Week 72
Change from baseline through Week 72 in Integrated Alzheimer's Disease Rating Scale (iADRS) | Baseline - Week 72
Change from baseline through Week 72 in Mini-Mental State Examination (MMSE) | Baseline - Week 72
Change from baseline in CDR-SB | Baseline up to but excluding Week 72
Time to increase in Clinical Dementia Rating, Global Score (CDR-GS) | Baseline - Week 72
Percentage of participants with adverse events (AEs) | Baseline - Week 72
Percentage of participants with amyloid-related imaging abnormalities (ARIA) magnetic resonance imaging (MRI) findings | Baseline - Week 72
Percentage of participants with infusion-related reactions (IRR) | Baseline - Week 72
Percentage of participants with anti-drug antibodies (ADAs) to trontinemab | Baseline - Week 72
Change from baseline through Week 72 in brain amyloid load as measured by amyloid positron emission tomography (PET) scan | Baseline - Week 72
Change from baseline to Week 72 in brain tau load as measured by tau PET scan in a subset of participants | Baseline - Week 72
Change from baseline through Week 72 in cerebrospinal fluid (CSF) biomarkers of disease p-tau181, neurogranin, Aβ42 in a subset of participants | Baseline - Week 72
Change from baseline through Week 72 in blood biomarkers p-tau217, glial fibrillar acidic protein (GFAP) | Baseline - Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (104):
- United States (26):
  - Banner Alzheimer?s Institute, Phoenix, Arizona
  - Healthy Brain Clinic, Long Beach, California
  - Oakland Clinical, Oakland, California
  - Riverside Clinical, Riverside, California
  - Cenexel California Neuroscience Research, LLC, Sherman Oaks, California
  - JEM Research LLC, Atlantis, Florida
  - K2 Medical Research-Winter Garden, Clermont, Florida
  - Visionary Investigators Network- Neurology Aventura, Miami, Florida
  - Charter Research - Winter Park/Orlando, Orlando, Florida
  - Conquest Research - Lake Nona, Orlando, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Great Lakes Clinical Trials Chicago d/b/a Flourish Research Andersonville, Chicago, Illinois
  - Adams Clinical Watertown, Watertown, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - Summit Research Network Inc., Portland, Oregon
  - Flourish Research ? Philadelphia, Plymouth Meeting, Pennsylvania
  - Gadolin Research, LLC, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Mt.Olympus Medical Research, Katy, Texas
  - Sana Research, LLC, Arlington, Virginia
  - Re:Cognition Health, Fairfax, Virginia
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Clinica Clinilive ltda, Maringá, Paraná, Brazil
- Canada (4):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Parkwood Institute Main Building, London, Ontario
  - The Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
- France (8):
  - CHU Amiens Hopital Sud, Amiens Cedex1
  - Centre Hospitalier Universitaire de Bordeaux Hopital Pellegrin, Bordeaux
  - Groupement Hospitalier Est - Hôpital Neurologique, Bron
  - CHU Dupruytren - Limoges, Limoges
  - Hopital Gui de Chauliac, Montpellier
  - Ch Pitie Salpetriere, Paris
  - CHU de Rouen Hopital, Rouen
  - Hop Guillaume Et Rene Laennec, Saint-Herblain
- Germany (13):
  - Ambulates Gesundheitszentrum der Charité GmbH, Berlin
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - German Center for Neurodegenerative Diseases (DZNE), Bonn
  - Universitätsklinikum Köln, Cologne
  - Medizinische Fakultät Carl Gustav Carus, Dresden
  - Universitätsklinikum des Saarlandes Klinik f. Psychiatrie und Psychotherapie, Homburg/Saar
  - Universitätsklinikum Jena, Klinik für Neurologie, Jena
  - Universität Leipzig, Leipzig
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Zentralinstitut für Seelische Gesundheit Abt.Gerontopsychiatrie, Mannheim
  - LMU Klinikum, Neurologische Klinik und Poliklinik, München
  - Ludwig-Maximilians-Univ., München
  - Universitätsklinikum Münster, Münster
- Ospedale Isola Tiberina - Gemelli Isola, Rome, Lazio, Italy
- Japan (9):
  - Brain Attack Center Ota Memorial Hospital, Hiroshima
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Kobe University Hospital, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Kochi Medical School Hospital, Kochi
  - Okayama City Hospital, Okayama
  - Rijikai Medical Corporation Katayama Medical Clinic, Okayama
  - Kotobuki Social Medical Corporation Tominaga Clinic, Osaka
  - Higashi-Shinjuku Clinic, Tokyo
- Poland (7):
  - O?rodek Badawczo-Naukowo-Dydaktyczny Chorób Ot?piennych w ?cinawie, ?cinawa
  - Uniwersytet Medyczny w Lodzi, ?ód?
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Medyczne "MEDYK", Rzeszów
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - NeuroProtect, Warsaw
- South Korea (11):
  - Pusan National University Hospital, Busan
  - Ajou University Medical Center, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Fundación ACE, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario la Fe, Valencia
- United Kingdom (10):
  - ReMind UK, Bath
  - Re:Cognition Health Birmingham, Birmingham
  - Scottish Brain Sciences, Edinburgh
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - St George?s Hospital, London
  - UCL Institute of Neurology, London
  - Manchester Mental Health and Social Care Trust, Manchester
  - Warneford Hospital, Oxford
  - Lancashire and South Cumbria NHS Foundation Trust, Preston
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing